CLINICAL TRIAL: NCT00664235
Title: Study of Thermal Imaging as an Objective RISK Indicator; The Evaluation of Skin Blood Flow and Temperature by Long Wave Infra-Red Imaging to Determine Effectiveness as a Predictor of Pressure Ulcer or Non-Visible Deep Tissue Damage
Brief Title: The Analysis of Skin Temperature by Long Wave Infrared Imaging to Determine Its Effectiveness as a Predictor of Tissue Injury
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Trillennium Medical Imaging, Inc. (Industry)
Responsible Party: Claude S. Burton, Professor of Medicine, Director Wound Management Institute, Duke University Medical Center
Other Study IDs: Pro00003228
Record Dates: First submitted 2008-04-21; First posted 2008-04-22 (Estimated); Last update posted 2008-04-22 (Estimated); Status verified 2008-04

CONDITIONS: Pressure Ulcers; Tissue Injury
Keywords: Pressure Ulcers; Tissue Injury
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Long-wave infrared imaging can be used to identify skin temperature changes associated with underlying tissue changes. We want to determine if the use of Long Wave infrared Imaging is as effective as the Braden Score in predicting nosocomial pressure ulcers.

DETAILED DESCRIPTION:
The Trillennium Medical Imaging system will be used to gather skin temperature data on 100 subjects. The subjects will be enrolled from Duke North floors 8100 or 8300 in a prospective controlled trial. All eligible patients who have signed a consent form will be assessed using the Long Wave Infrared imaging.

Subjects eligible for this study who have signed a consent form will be scanned on bilateral heels and sacrum. Subjects with ulcers on those areas will also be scanned due to the fact that they are at a high risk of developing additional pressure ulcers. The intent is not to capture images of the existing ulcer, but to focus on areas that could potentially develop into additional pressure ulcers. The subjects who already have an ulcer will only be scanned on non ulcerated tissue. The areas of interest must be off-loaded for 3 minutes from any pressure in order to acclimate to ambient temperature. The device will be held approximately 36 inches from the area of interest in order to obtain an image. The subjects will be assessed within 24 hours of admission and every 24 hours until discharge or they develop a pressure ulcer. The subject's routinely recorded Braden scores (By on the floor nursing staff) will also be captured in order to effectively compare the effectiveness of the Imaging system. The nurse conducting the imaging will also record a Braden score.

All subjects will be included in the trial unless they refuse to participate or are incapacitated to the degree that imaging becomes unreasonable.

ELIGIBILITY:
Inclusion Criteria:

* To be admitted to 8100 or 8300 and be willing to participate in the study

Exclusion Criteria:

* Unwillingness to participate

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients will be recruited from Duke North inpatient unit 8100 or 8300. All patients admitted to the above floor will be evaluated for willingness to participate.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2008-02; Primary Completion 2008-04 (Estimated); Study Completion 2008-06 (Estimated)

PRIMARY OUTCOMES:
Each time a pattern of injury is identified by the device, we will correlate this occurrence with the Braden scale to see whether or not it suggested an injury potential. | 90 days

SECONDARY OUTCOMES:
It is our hypothesis that the pattern of injury will develop without warning from the Braden scores. | 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Claude S. Burton, M.D., Principal Investigator — Duke Health
Locations (1):
- Duke University Health System, Durham, North Carolina, United States